CLINICAL TRIAL: NCT03130049
Title: The Effect of the Popliteal Plexus Block on Postoperative Pain After Reconstruction of the Anterior Cruciate Ligament
Brief Title: Popliteal Plexus Block for Postoperative Pain After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protokol_PPB_ACL_21042017
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-04

CONDITIONS: Anterior Cruciate Ligament Injury; Postoperative Pain
Keywords: Peripheral nerve block; Ultrasound
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with postoperative pain, NRS >3 (Experimental): Patients reporting postoperative pain (NRS >3) localized to the center of the knee (10 patients) will receive a popliteal plexus block
  Interventions: Procedure: Popliteal plexus block
- Patients with postoperative pain, NRS ≤ 3 (No Intervention): (approx. 90 patients)

INTERVENTIONS:
Procedure: Popliteal plexus block — 10 mL Marcain-adrenalin 5 mg/mL + 5 microgram/mL. Ultrasound-guided injection into the distal part of the adductor canal
  Arms: Patients with postoperative pain, NRS >3

SUMMARY:
The study aims to investigate the effect of the popliteal plexus block (PPB) on postoperative pain in patients undergoing anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
Postoperative pain following ACL reconstruction can be alleviated with an ultrasound-guided femoral triangle block (FTB). However, it is the investigators' observation that 10-20 % of the patients still complain of intense pain localized in the center of the knee.

Cadaver dissection studies have shown that an injection into the distal part of the adductor canal will spread to the popliteal fossa, and one dissection study showed consistent spread to the popliteal plexus.

The study team hypothesized that a PPB will reduce the postoperative pain, when it is used as a supplement to the FTB in patients undergoing ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL reconstruction on one of the two trial sites
* Age ≥ 18
* American Society of Anesthesiologists (ASA) status I-III
* Informed consent

Exclusion Criteria:

* Patients unable to cooperate
* Patients not able to speak Danish or with other communication problems
* Pregnancy
* Contraindication towards any medical product used in the study
* Preoperatively reduced sensation on the medial and lateral part of the lower leg
* Patients with diabetes requiring medical treatment
* Preoperative intake of opioids (dosed > once daily)
* ACL revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
The effect of the popliteal plexus block (PPB) | Pain scores (NRS): 15, 30, 45 and 60 minutes after PPB
  Evaluated as the percentage of patients with postoperative pain NRS >3, dropping in pain score to NRS ≤ 3 after the PPB

SECONDARY OUTCOMES:
Percentage of patients with central knee pain | Pain scores: 15, 30, 45 and 60 minutes after arrival at the post anesthesia care unit (PACU)
  The percentage of patients with FTB reporting pain (NRS >3) localized in the center of the knee in the observation period
Onset time for PPB | Pain scores (NRS): 15, 30, 45 and 60 minutes after PPB
  Time from withdrawal of the needle until patient reports NRS ≤ 3
The effect of the PPB on cutaneous sensation | Baseline, 30 and 60 minutes after PPB
  Tested on the lateral part of the lower leg (pinprick test)
The effect of the PPB on muscle strength | Baseline, 60 minutes after PPB
  Dorsal flexion and plantar flexion in the ankle joint, measured with a handheld dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Jensen, MD, Principal Investigator — Aarhus University Hospital; Christian Jessen, MD, Principal Investigator — The Regional Hospital in Horsens
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus C
  - The Regional Hospital in Horsens, Horsens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wong WY, Bjorn S, Strid JM, Borglum J, Bendtsen TF. Defining the Location of the Adductor Canal Using Ultrasound. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):241-245. doi: 10.1097/AAP.0000000000000539. PMID 28002228
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Background] Goffin P, Lecoq JP, Ninane V, Brichant JF, Sala-Blanch X, Gautier PE, Bonnet P, Carlier A, Hadzic A. Interfascial Spread of Injectate After Adductor Canal Injection in Fresh Human Cadavers. Anesth Analg. 2016 Aug;123(2):501-3. doi: 10.1213/ANE.0000000000001441. PMID 27442773